CLINICAL TRIAL: NCT00611377
Title: Delirium in Patients Admitted to a Respiratory Weaning Centre: Analysis of Incidence and Risk Factor
Brief Title: Study on the Incidence of Delirium in a Respiratory Weaning Centre
Acronym: delricu
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Piero Ceriana, Fondazione Salvatore Maugeri
Other Study IDs: delirium in rwc; deliriumPavia
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-01

CONDITIONS: Delirium
Keywords: delirium; mechanical ventilation; age; severity score
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
Delirium is rather common among patients in Intensive Care Units (ICU), while little is known about its incidence in ventilator-dependent patients transferred to a Weaning Center (WC), once in a phase of clinical stability. We will prospectively evaluate for the presence of delirium all the ventilator-dependent patients admitted to our WC over a period of two years. They will be monitored using the Intensive Care Delirium Screening Checklist (ICDSC), previously validated in the ICU setting. This evaluation is based on a score based on 8 items obtained with a simple examination by the attending physician. The final sum generates a score considered normal (0-1), borderline (2-3) and pathologic (>4). All the patients, except those with normal score, will also be evaluated by a psychiatrist, using the Diagnostic Manual of Mental Disorders (DSM-IV), considered the gold standard. The score will be assessed at patient's admission, at mid-hospital stay and at discharge.

DETAILED DESCRIPTION:
Delirium has been defined, according to the Diagnostic and Statistical Manual of Mental Disorders (DSM IV), as a disturbance of consciousness characterized by an acute onset and fluctuating course. This impairment of cognitive functions, not being accounted for by a pre-existing dementia, reduces the patient's ability to receive, process and recall informations and its main features are inattention, disorganized thinking and reduced clarity of awareness of the environment.

All patients transferred from an intensive care unit to our respiratory weaning centre (RWC) will be screened for the occurrence of delirium. Our RWC is a 7-bed unit located within the respiratory department of a rehabilitation hospital and is fully equipped for invasive and non-invasive mechanical ventilation (MV) and for invasive and noninvasive cardiorespiratory monitoring. Patients are generally transferred to our unit from a general or surgical ICU for weaning from MV or, in case of patients already weaned, for rehabilitation, monitoring and intensive nursing care. All patients or their next of kin will give written informed consent to participate to the study and the study protocol has been approved by the local ethics committee.

For the assessment of delirium we use the Intensive Care Delirium Screening Checklist (ICDSC),a diagnostic tool already validated in the intensive care setting even in mechanically ventilated patients. It is based on the assessment of 8 different items dealing with the patient's mental status: each one is scored 0 or 1 in case of, respectively, absence or presence of the item itself and the final score is the resultant of the sum of the different items (see the appendix 1 for further details). The evaluation is performed on a daily basis by the physician in charge and the ICDSC score is ranked in the following way: 0 to 1 is considered normal, 2 to 3 is considered borderline, (i.e. indicative of a subsyndromal delirious state) and 4 or greater is considered diagnostic for delirium (13). In presence of a score greater than 1 the psychiatrist is called for consultation and diagnostic confirmation. Upon discharge of the patient from our RWC a score trend is drawn for every patient using the three highest scores sampled during the phases of admission, of mid stay and of discharge. Cases of overt delirium (only patients with ICDSC score ≥4) are categorized as hyperactive or hypoactive, according to a currently accepted classification. Treatment of delirium, when properly diagnosed, is instituted according to the psychiatist's prescriptions.

Patient's data collection include demographic data (age, gender), severity score (SAPS II), reason for admission (i.e. need for mechanical ventilation (MV) or not (NMV)) and previous episodes of delirium (hyperactive forms) occurring during ICU stay not linked to a pre-existing mental disease or to an acquired brain failure of vascular, metabolic or infectious origin. The Kelly scale is used for the assessment of the level of consciousness: the patient is considered comatose in presence of a persistent (>24 hours) Kelly score of ≥4. As far as the use of sedatives and analgesics in our RWC is concerned, our policy is based on the avoidance of continuous infusions regimens and on the limitation to the use of those drugs with a known or suspected capability to induce delirium; each drug is prescribed when strictly needed according to the judgement of the physician on duty and is targeted to the treatment of the specific symptom: pain, anxiety, insomnia etc.

Analysis of variance for repeated measures (MANOVA) is employed for statistical analysis, and a p value lower than 0.05 is considered the threshold value for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted in the respiratory weaning centre

Exclusion Criteria:

* Patients in deep coma
* Deceased or transferred to another ward within 72 hours of admission

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will evaluate for the presence of delirium all the ventilator-dependent patients admitted to our RWC. They will be monitored using the Intensive Care Delirium Screening Checklist (ICDSC). This evaluation is based on a score based on 8 items obtained with a simple examination by the attending physician. The final sum generates a score considered normal (0-1), borderline (2-3) and pathologic (>4). All the patients, except those with normal score, will also be evaluated by a psychiatrist, using the Diagnostic Manual of Mental Disorders (DSM-IV), considered the gold standard. The score will be assessed at patient's admission, at mid-hospital stay and at discharge.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-02 (Estimated); Study Completion 2008-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Piero M Ceriana, Principal Investigator — Fondazione Salvatore Maugeri
Locations (1):
- Department of respiratory medicine and intensive care unit, Pavia, PV, Italy